CLINICAL TRIAL: NCT00510380
Title: Epigenetic Markets in Growth Restricted Human Pregnancies: A Case- Control Study
Brief Title: Epigenetic Markers in Growth Restricted Human Pregnancies: a Case-controlled Study
Status: Completed | Type: Observational
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Chong Yap Seng, National University Hospital, Singapore
Other Study IDs: SIG/07072
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Last update posted 2009-09-21 (Estimated); Status verified 2009-09

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- growth-restricted Chinese pregnancies
- appropriately-grown Chinese pregnancies

SUMMARY:
This study is carried out to discover if a baby with restricted growth in the womb is subject to specific fetal programming which predisposes to the metabolic syndrome(diabetes,hypertension,heart disease) in adulthood.We have elected to first study this condition in Chinese population in Singapore with the eventual plan of studying all ethnic groups. This is important for understanding the molecular basis of adult-onset disease such as diabetes, identifying children at risk of developing this disease in future and targeting specific strategies for intervention and disease prevention.

Intrauterine fetal programming is effected through epigenetic changes similar to those previously identified in animal studies. The epigenetic markers can be found in growth restricted Chinese pregnancies in the local population.

DETAILED DESCRIPTION:
Fetal growth restriction is associated with accelerated postnatal weight gain and increased obesity risk in later life.International epidemiological data suggest that the phenomenon of fetal programming links poor intrauterine growth to adult disease, primarily type II diabetes, obesity and metabolic syndrome, conditions increasingly common in Singapore. Suboptimal intrauterine environmental condition s are postulated to affect fetal development through effects on developmental plasticity through epigenetic processes. These effects manifest as poor glucose resistance, insulin resistance, obesity and cardiovascular disease in later life. There is increasing animal data to support this model.

The aim of this study is to determine if epigenetic markers of the metabolic syndrome are present in selected Chinese pregnancies in Singapore.

Hypothesis:

Intrauterine fetal programming is effected through epigenetic changes similar to those previously identified in animal studies. The epigenetic markers can be found in growth restricted Chinese pregnancies in the local population.

Methodology Umbilical cords and cord blood will be collected from twenty unequivocally growth-restricted Chinese pregnancies and twenty appropriately-grown Chinese pregnancies. DNA extracted from these tissues will be subjected to a custom-made DNA methylation array probing for specific changes in 262 candidate genes important to fetal endocrine and metabolic control.

This will be done using either a methylation array or a Sequenorn 2 in the DNA extracts that have been identified through Epigen academic consortium of the Liggins Institute and UK collaborators.

Anthropometric data will be collected from the infants at birth, and subsequently at 3,6,12,18 and 24 months and we will seek differential measures of programming.

Application The discovery of biomarkers indicating shifted developmental trajectories is the most important need in developmental programming research. Birth weight alone is not a valid measure. Biomarkers predictive of later obesity and the metabolic syndrome will be invaluable in formulating preventive strategies for these diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese women,
2. Singleton pregnancies,
3. fetal growth restriction diagnosed clinically and by ultrasound parameters,
4. Normally grown fetuses by clinical and ultrasound criteria

Exclusion Criteria:

1. Non-Chinese women
2. Multiple pregnancies
3. Co-existing antenatal complications including sever pre-eclampsia

Ages: 21 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Babies from Chinese women with single pregnancies
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2007-04; Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yap Seng Chong, MBBS, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Hospital, Singapore, Singapore